CLINICAL TRIAL: NCT03775837
Title: Effect of Panax Ginseng C.A. Mey Extract on Liver Function in Adults: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Panax Ginseng C.A. Mey Extract on Liver Function in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2018-031
Record Dates: First submitted 2018-12-11; First posted 2018-12-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Panax Ginseng C.A. Mey Extract group (Experimental): This group takes Panax Ginseng C.A. Mey Extract for 8 weeks
  Interventions: Dietary Supplement: Panax Ginseng C.A. Mey Extract group
- Placebo group (Placebo Comparator): This group takes placebo for 8 weeks
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Panax Ginseng C.A. Mey Extract group — This group takes Panax Ginseng C.A. Mey Extract for 8 weeks
  Arms: Panax Ginseng C.A. Mey Extract group
Dietary Supplement: Placebo group — This group takes placebo for 8 weeks
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Panax Ginseng C.A. Mey Extract on liver function in adults for 8 weeks.

DETAILED DESCRIPTION:
Previous studies have indicated that Panax Ginseng C.A. Mey Extract may have the ability to improve liver function. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of the Panax Ginseng C.A. Mey Extract on liver function in adults; the safety of the compound are also evaluate. The Investigators examine AST, ALT, GGT, and other metabolic parameters at baseline, as well as after 4 and 8 weeks of intervention. Sixty adults were administered either 600 mg of Panax Ginseng C.A. Mey Extract or a placebo each day for 8 weeks;

ELIGIBILITY:
Inclusion Criteria:

* ALT ranging from upper limit of reference to three times of upper limit

Exclusion Criteria:

* Abnormal liver or renal function (i.e., serum aminotransferase activity > 3 times of upper limit of reference range and serum creatinine concentrations > 1.2 mg/dL)
* Diabetes (diagnosed clinically or fasting glucose level > 126 mg/dL)
* History of viral hepatitis or cancer
* Uncontrolled hypertension
* History of serious cardiac disease such as angina or myocardial infarction
* History of gastrectomy
* History of medication for psychiatric disease
* Administration of oriental medicine including herbs within the past 4 weeks

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Alanine aminotransferase | 8 weeks
  Alanine aminotransferase

SECONDARY OUTCOMES:
Aspartate aminotransferase | 8 weeks
  Aspartate aminotransferase
Gamma-glutamyl transferase | 8 weeks
  Gamma-glutamyl transferase

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Integrated Research Institute for Natural Ingredients and Functional Foods, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No